CLINICAL TRIAL: NCT03665467
Title: The Global Prevalence of Infections in Urology Study
Acronym: GPIU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Association of Urology Research Foundation (Other)
Responsible Party: Principal Investigator, Florian M E Wagenlehner, Professor of Urology, University of Giessen
Other Study IDs: GPIU
Record Dates: First submitted 2018-07-08; First posted 2018-09-11 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hospital Infection; Urinary Tract Infections
MeSH Terms: conditions — Cross Infection; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urology departments from all over the world are invited to join the Global Prevalence Study on Infections in Urology (GPIU-study) and the GPIU Prostate Biopsy Side Study. The GPIU study is taking part annually in November since 2003. European urologists were the first group of specialist to register hospital acquired infections on an international level. More than 20.000 patients have been screened and more than 2000 patients are currently listed in this database.

Why? Infectious complications after urological procedures, such as prostate biopsy and increasing antimicrobial resistance are posing significant threats to modern urology The GPIU-study is a combined quality improvement initiative and a scientific study. Once the participating departments have filled in the report forms they will get access to statistics showing the accumulated results for all participating hospitals. The participants can anonymously compare their own results with hospitals from all over the World. The GPIU-study application has been designed as an instrument to ongoing follow-up of the development of important factors related to infection on international, national and local levels.

Take responsibility for the future of urology - join the GPIU-studies! http://gpiu.esiu.org

Prof. Dr. Florian M.E. Wagenlehner, MD, PhD Clinic for Urology, Pediatric Urology and Andrology University Clinic Giessen, Germany GPIU study coordinator

Prof. Truls E. Bjerklund Johansen, MD, PhD Urology Department, Oslo University Hospital, Chairman ESIU Oslo, NO GPIU Study coordinator

Zafer Tandogdu University College London (UCL), UK

Dominic Althaus Software engineer Giessen, Ger

ELIGIBILITY:
* On the chosen single study day at 08:00 AM local time all patients present on the ward of the participating institution are included
* The presence of urinary tract infections (UTI) according to the CDC definitions during their entire hospital stay are documented and audited and the patients are categorized as having or not having a UTI and/or
* The presence of surgical site infection (SSI) according to the CDC definitions during their entire hospital stay are documented and audited and the patients are categorized as having or not having a SSI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -hospitalised urological patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-11-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Health care associated infection episode | an infection onset 48 hours after admission to hospital or after an intervention
  Health Care Associated Infections per definition of the Center for Disease Control

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wagenlehner, Prof., Study Chair — Giessen University; Zafer Tandogdu, Principal Investigator — Mr; Truls Erik Bjerklund Johansen, Prof., Study Director — Oslo University; Bela Koves, PhD, Principal Investigator — Jahn Ferenc South Pest Teaching Hospital
Locations (4):
- Giessen University, Medical School, Giessen, Germany
- Jahn Ferenc South Pest Teaching Hospital, Budapest, Hungary
- Oslo University, Oslo, Norway
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
* Investigators will be able to download their own submitted data
  * Investigators will be able to access an online summary statistics of the annual pooled sample
  * Investigators will be able to compare their own summary statistics with other centers on the study website.
Supporting Information: Study Protocol, CSR
Time Frame: Annual
Access Criteria: Study investigators will be able to access their own data and in addition the summary statistics of the pooled sample on an annual basis.
URL: http://gpiu.esiu.org/

REFERENCES:
- [Background] Wagenlehner F, Tandogdu Z, Bartoletti R, Cai T, Cek M, Kulchavenya E, Koves B, Naber K, Perepanova T, Tenke P, Wullt B, Bogenhard F, Johansen TE. The Global Prevalence of Infections in Urology Study: A Long-Term, Worldwide Surveillance Study on Urological Infections. Pathogens. 2016 Jan 19;5(1):10. doi: 10.3390/pathogens5010010. PMID 26797640
- [Background] Wagenlehner F, Tandogdu Z, Bartoletti R, Cai T, Cek M, Kulchavenya E, Koves B, Naber K, Perepanova T, Tenke P, Wullt B, Bogenhard F, Bjerklund Johansen TE; GPIU Investigators. The Global Prevalence of Infections in Urology (GPUI) Study: A Worldwide Surveillance Study in Urology Patients. Eur Urol Focus. 2016 Oct;2(4):345-347. doi: 10.1016/j.euf.2016.03.004. Epub 2016 Apr 1. PMID 28723463
- [Background] Tandogdu Z, Bartoletti R, Cai T, Cek M, Grabe M, Kulchavenya E, Koves B, Menon V, Naber K, Perepanova T, Tenke P, Wullt B, Johansen TE, Wagenlehner F. Antimicrobial resistance in urosepsis: outcomes from the multinational, multicenter global prevalence of infections in urology (GPIU) study 2003-2013. World J Urol. 2016 Aug;34(8):1193-200. doi: 10.1007/s00345-015-1722-1. Epub 2015 Dec 11. PMID 26658886
- [Background] Cek M, Tandogdu Z, Wagenlehner F, Tenke P, Naber K, Bjerklund-Johansen TE. Healthcare-associated urinary tract infections in hospitalized urological patients--a global perspective: results from the GPIU studies 2003-2010. World J Urol. 2014 Dec;32(6):1587-94. doi: 10.1007/s00345-013-1218-9. Epub 2014 Jan 23. PMID 24452449
- [Background] Tandogdu Z, Cek M, Wagenlehner F, Naber K, Tenke P, van Ostrum E, Johansen TB. Resistance patterns of nosocomial urinary tract infections in urology departments: 8-year results of the global prevalence of infections in urology study. World J Urol. 2014 Jun;32(3):791-801. doi: 10.1007/s00345-013-1154-8. Epub 2013 Aug 24. PMID 23979151
- [Background] Cek M, Tandogdu Z, Naber K, Tenke P, Wagenlehner F, van Oostrum E, Kristensen B, Bjerklund Johansen TE; Global Prevalence Study of Infections in Urology Investigators. Antibiotic prophylaxis in urology departments, 2005-2010. Eur Urol. 2013 Feb;63(2):386-94. doi: 10.1016/j.eururo.2012.09.038. Epub 2012 Sep 25. PMID 23031676
- [Background] Wagenlehner FM, van Oostrum E, Tenke P, Tandogdu Z, Cek M, Grabe M, Wullt B, Pickard R, Naber KG, Pilatz A, Weidner W, Bjerklund-Johansen TE; GPIU investigators. Infective complications after prostate biopsy: outcome of the Global Prevalence Study of Infections in Urology (GPIU) 2010 and 2011, a prospective multinational multicentre prostate biopsy study. Eur Urol. 2013 Mar;63(3):521-7. doi: 10.1016/j.eururo.2012.06.003. Epub 2012 Jun 12. PMID 22704727